CLINICAL TRIAL: NCT03460184
Title: Effect of Different Types of Anesthesia on Perioperative Brain Natriuretic Peptide Levels in Parturient Cardiac Patient Undergoing Elective Cesarean Section
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Sahr Marzouk (Unknown); Heba Omar (Unknown); Michael Wahib Wadeed (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Other Study IDs: N-2-2018
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: General Anesthesia Versus Spinal Anesthesia on BNP Hormone Levels Preoperatively and Postoperatively in Parturient Cardiac Patient Undergoing C.S

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- G.A Group A: Group A: n= 30 Parturiant patients will receive general anesthesia. General anesthesia will be conducted After pre-oxygenation for 3-5 minutes. 5% thiopental (5 mg/kg) will be administered intravenously over 30s, followed by succinylcholine 1.5 mg/kg. After tracheal intubation, the patients will be ventilated with 100% oxygen. isoflurane 0.8% will be added, to maintain the anesthesia. Further neuromuscular block will be maintained by using atracurium as needed. After delivery of the fetus, fentanyl IV will be given 1ug/kg as analgesia and 20 IU oxytocin will be given by intravenous infusion .Reverse neuromuscular blockade as necessary at completion of surgery. Extubate when the patient is awake, the anesthesia is adequately reversed, and the patient is following commands
  Interventions: Diagnostic Test: G.A Group A:
- Spinal A Group B: Group B: n= 30 Parturiant patients will receive spinal anesthesia. In the sitting position and after complete aseptic precaution are taken, 2-3 ml of Lidocaine will be injected subcutaneously, spinal anesthesia will be performed at interspace L3-4 or L4-5, either via midline or paramedian approaches using 22 guage Quinke needle with the bevel directed laterally. 2.5 ml of hyperbaric bupivacaine 0.5% in addition to 25 μg fentanyl (0.5 ml) will be injected into the subarachnoid space after successful dural puncture and confirmation by barbotage.
  The patient will be put flat in the supine position with left uterine displacement using wedge under the right loin and the surgeon will be allowed to sterilize and wrap the field after confirmation of the solidity of the block its level.
  All patiens will be observed for cardiac complications in the form of non-fatal MI, arrhythmias and sudden cardiac death until discharged after at least 72h.
  Interventions: Diagnostic Test: G.A Group A:

INTERVENTIONS:
Diagnostic Test: G.A Group A: — G.A will be conducted After pre-oxygenation for 3-5 minutes. thiopental (5 mg/kg) will be administered I.V, followed by succinylcholine 1.5 mg/kg. After tracheal intubation, the patients will be ventilated with 100% oxygen. isoflurane 0.8% will be added, to maintain the anesthesia. Further neuromuscular block will be maintained by using atracurium . After delivery of the fetus, fentanyl IV will be given 1ug/kg as analgesia and 20 IU oxytocin will be given by I.V infusion .Reverse neuromuscular blockade as necessary at completion of surgery. Extubate when the patient is awake
  In the sitting position and after complete asepsis , 2-3 ml of Lidocaine will be injected subcutaneously, spinal anesthesia will be performed at interspace L3-4 or L4-5, midline approaches using 22 guage Quinke needle . 2.5 ml of hyperbaric bupivacaine 0.5% in addition to 25 μg fentanyl will be injected into the subarachnoid space after successful dural puncture and confirmation by barbotage.
  Other Names: Spinal A Group B:

SUMMARY:
comparing the effect of general anesthesia versus spinal anesthesia on brain natruretic peptide hormone levels preoperatively and postoperatively in parturient cardiac patient undergoing cesarean section

DETAILED DESCRIPTION:
In our study, investigators will detect changes in brain natruretic peptide (BNP) levels in parturient patients at risk undergoing cesarean section, in relation to type of anesthesia used, general anesthesia versus spinal anesthesia, in order to evaluate the safety of type of anesthesia used for this kind of patient.

It is very important to assess and predict risk in the cardiovascular system in such cases. A number of cardiac indexes for predicting risk have been developed like Goldman Multifactorial risk index, Eagle's risk index and Detsky's cardiac index. It is recommended to evaluate patients using these indexes and to institute preoperative medical treatment based on the results. These clinical scoring systems, although simple to use, are somewhat inconvenient and have limitations in their predictive value, whereas other cardiac investigations such as exercise or pharmacologic stress imaging are sensitive, but limited in practice by time and resources. Recently brain natriuretic peptide (BNP) was spotlighted as a predictor for diagnosing and predicting the prognosis of various heart diseases. BNP is a cardiac hormone that is synthesized by ventricular myocytes in response to ventricular dysfunction. Recent studies have demonstrated that elevated serum BNP levels predict first cardiovascular event and death in the general population. In addition, it has been reported that BNP measured before major surgery can be used as a predictor of postoperative cardiac complications.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate valvular heart lesions.
* Cardiomyopathic lesions with ejection fraction > 40%
* Ischemic heart disease
* Hypertension
* Non-fatal arrhythmias eg. Controlled AF

Exclusion Criteria:

Cardiomyopathic lesions with EF less than 40% Tight stenotic lesions Severe regurgitant lesions Pregnancy induced hypertension Fatal arrhythmia eg. Ventricular tachycardia renal impairment Cr > 1.2 surgery related problems: operation longer than 3 hours patient resuscitation with > 3 litres blood loss more than 1 liter

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturient cardiac patient undergoing cesarean section.
Study Population: Parturient cardiac patient 20-50 years old undergoing cesarean section with
  * Mild to moderate valvular heart lesions.
  * Cardiomyopathic lesions with ejection fraction > 40%
  * Ischemic heart disease
  * Hypertension
  * Non-fatal arrhythmias eg. Controlled AF
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Monitoring changes in BNP | 24 hours postoperative
  Monitoring changes in BNP level pre and postoperatively in relation to type of anesthesia to evaluate the safety of type of anesthesia used in cesarean section for parturient with cardiac diseas

SECONDARY OUTCOMES:
Hemodynamic monitoring | 24 hours postoperative
  Monitor changes in hemodynamics in relation to type of anesthesiaM
Efficiency of BNP | 24 hours postoperative
  Efficiency of BNP in detection of cardiac complications

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Population of study & disease condition Following ethical committee approval, the study will be carried out on 30 parturient patients with cardiac disease undergoing cesarian section at Kasr El Ainy hospitals after obtaining the informed consent.